CLINICAL TRIAL: NCT06805006
Title: i-Stitch for Bilateral Sacrospinous Ligament Fixation (SSLF)
Acronym: i-StitchSSLF
Status: Enrolling by invitation | Type: Observational
Sponsor: A.M.I. Agency for Medical Innovations GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: PMCF-03-011
Record Dates: First submitted 2025-01-28; First posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Pelvic Organ Prolapse; Genital Prolapse
Keywords: bilateral sacrospinous ligament fixation; suture attachment medical device
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: SSLF — Bilateral sacrospinous ligament fixation with i-Stitch device

SUMMARY:
The purpose of the clinical investigation is to generate clinical data to substantiate the safety and performance of the i-Stitch device for bilateral sacrospinous ligament fixation (SSLF) in pelvic organ prolapse (POP) repair.

DETAILED DESCRIPTION:
The i-Stitch instrument is a reusable instrument for attaching sutures to tissue with or without surgical mesh implants in urogynaecology. It is used together with the i-Stitch loading units. The use of i-Stitch for the fixation of surgical urogynaecological mesh implants (e.g. BSC Mesh, InGYNious) has already been proven in several studies.

The aim of the present retrospective study is to generate clinical data to show the safety and performance of the i-Stitch instrument in bilateral sacrospinous ligament fixation (SSLF) without the use of a surgical mesh.

ELIGIBILITY:
Inclusion Criteria:

* Surgery for POP
* SSLF with usage of i-Stitch device (& i-Stitch Loading Units)
* Concomitant procedures are allowed
* Women minimum 18 years old
* Written informed consent for surgery

Exclusion Criteria:

* infection (active or latent)
* allergies to the materials used
* benign or malignant changes
* anticoagulation disorders
* autoimmune connective tissue disorders
* any uterus pathologies

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients with symptomatic pelvic organ prolapse indicated for a surgical intervention.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Subjective outcome | 12 months
  German Pelvic Floor Questionnaire ("Deutscher Beckenboden-Fragebogen")
Subjective outcome | 3 months
  German Pelvic Floor Questionnaire ("Deutscher Beckenboden-Fragebogen")

SECONDARY OUTCOMES:
Quality of life (ICIQ-UI SF) | 12 months
  urinary incontinence and its impact on quality of life using the short form of the International Consultation on Incontinence Questionnaire
Postoperative complications | 12 months
  Complications in women undergoing bilateral SSLF using the i-Stitch
Anatomical outcome (POP-Q) | 12 months
  Objective anatomical failure/recurrent prolapse in any anatomical compartment

CONTACTS AND LOCATIONS:
Overall Officials: Ursula Peschers, Prof. Dr., Principal Investigator — ISAR Klinikum Munich
Locations (1):
- Isar Kliniken GmbH, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No